CLINICAL TRIAL: NCT06342466
Title: A Study of Bortezomib, Pomalidomide, Dexamethasone in Patients with Systemic AL Amyloidosis
Brief Title: Bortezomib, Pomalidomide, Dexamethasone for Systemic AL Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jin Lu, MD (Other)
Responsible Party: Sponsor-Investigator, Jin Lu, MD, Principle Investigator, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-358-02
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-05

CONDITIONS: Systemic Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Bortezomib, pomalidomide, dexamethasone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BPd (Experimental): BPd regimen (Bortezomib, pomalidomide, and dexamethasone) will be applied every 28 days until progression of disease, unacceptable toxicity or subsequent therapy, for a maximum of six cycles.
  Interventions: Drug: Bortezomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3mg/m2 sc weekly
  Other Names: Velcade
Drug: Pomalidomide — 4mg per day taken orally on 1-21 of repeated 28-day cycles
Drug: Dexamethasone — Dexamethasone 20mg-40mg weekly

SUMMARY:
This is an open-label, multicenter, Phase 2 study in subjects with newly diagnosed or previous treated systemic light chain (AL) amyloidosis. Approximately 40 subjects will receive therapy with bortezomib, pomalidomide, and dexamethasone. The primary outcome is hematologic very good partial response and complete response rate at 6 months.

DETAILED DESCRIPTION:
Proteasome inhibitor and immunmodulators have synergistic effect for plasma cell dyscrasia. Due to the fact that more than 70-80% of patients with amyloidosis have renal involvement, the application of lenalidomide is limited. Thus, the investigators designed this open-label, multicenter, phase 2 study for newly diagnosed or previously treated systemic AL amyloidosis with bortezomib, pomalidomide and dexamethasone regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AL amyloidosis, confirmed by histology and typed with immunohistochemistry, immunoelectron microscopy or mass spectrometry.
2. Newly diagnosed or previous treated AL amyloidosis
3. Patients must be ≥ 18 years of age.
4. ECOG performance status 0, 1 or 2.
5. Measurable disease defined by at least one of the following:

   ① serum free light chain (FLC) ≥2.0 mg/dL (20 mg/L) with an abnormal kappa:lambda ratio or the difference between involved and uninvolved free light chains (dFLC) ≥2mg/dL (20 mg/L).

   ②. presence of a monoclonal spike that is ≥5 g/l.
6. Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system).
7. Absolute neutrophil count (ANC) ≥1.0 X 10^9/L, Hemoglobin ≥70 g/L, Platelets ≥50 X 10^9/L
8. eGFR ≥20 mL/min/ 1.73 m^2
9. Written informed consent in accordance with local and institutional guidelines.
10. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma.
2. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
3. Severe or persistent infection that cannot be effectively controlled;
4. Presence of severe autoimmune diseases or immunodeficiency disease;
5. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]);
6. Patients with HIV infection or syphilis infection;
7. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hematologic VGPR + CR rate at 6 months | 6 months
  Hematologic very good partial response plus complete response rate at 6 months

SECONDARY OUTCOMES:
Overall Hematologic response rate at 6 months | 6 months
  Overall Hematologic partial response, very good partial response rate and complete response at 6 months
At least one organ response at 6 months | 6 months
  At least one organ response (cardiac response, renal response, liver response) at 6 months
TTNT at 2 years | 2 years
  Time to next treatment at 2 years
Estimated PFS at 2 years | 2 years
  Estimated Progression free survival at 2 years
Estimated OS at 2 years | 2 years
  Estimated Overall Survival at 2 years
TRAE | 6 months
  Treatment-related adverse events up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No